CLINICAL TRIAL: NCT06917807
Title: Comparative Evaluation of Analgesic Efficacy of Ultrasound Guided Pericapsular Nerve Group Block and Quadratus Lumborum Block During Positioning of Patients With Proximal Femur Fractures for Spinal Anesthesia
Brief Title: Pain Relief Comparison: Pericapsular Nerve Group Versus Quadratus Lumborum Block for Positioning in Femur Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD02/2024/2025
Record Dates: First submitted 2025-03-06; First posted 2025-04-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Post Operative Pain; Hip Fracture; Regional Anaesthesia; Quadratus Lumborum Block
Keywords: regional anesthesia; pain managment; QLB block; PENG block; Hip fracture; postoperative analgesia; nerve block; opioid sparing anesthesia; acute pain control; clinical trial
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nervegroup block (Active Comparator): the regional block will be performed with the patient in the supine position. Ultrasound machine with low frequency curvilinear probe (2-5MHz) covered with sterile sheath will be initially placed in a transverse plane over the Anterior Inferior Iliac Spine (AIIS) and then aligned with the pubic ramus by rotating the probe counter-clockwise approximately 45 degrees. In this view, the Iliopectineal Eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A 22-gauge, 80-mm needle will be inserted from lateral to medial to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anaesthetic solution (30ml of bupivacaine 0.25%) will be injected in 5-mL increments while observing for adequate fluid spread in this plane, without exceeding the toxic dose (3 mg/kg)
  Interventions: Procedure: Pericapsuler nerve group block
- Quadratus lumborum block (Active Comparator): the block will be performed with the patient in the supine position. Under ultrasound guidance with a low frequency curvilinear probe (2-5MHz) covered with sterile sheath, the prob will be placed in coronal plane at midaxillary line between subcostal margin and iliac crest. A 22-gauge, 80-mm needle will be inserted distal to subcostal margin and advanced under curvilinear probe. The needle will be advanced through external oblique aponeurosis, internal oblique, and transversus abdominis muscles. Visualizing the tip penetrating the posterior epimysium of QLM and entering anterior thoracolumbar fascia (ATLF). A small volume of local anaesthetic will be injected after locating the needle tip and a negative aspiration for blood. After the distribution of the local anesthetic will be seen, the rest of the 30 mL of 0.25 % of bupivacaine will be injected
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Pericapsuler nerve group block — A single shot pericapsular nerve group block preformed under ultrasound guidance with a local anesthetic agent ( Marcaine )
  Arms: Pericapsular nervegroup block
Procedure: Quadratus lumborum block — A single shot Quadratus lumborum block preformed under ultrasound guidance with a local anesthetic agent ( Marcaine )
  Arms: Quadratus lumborum block

SUMMARY:
This study aims to compare the analgesic efficacy of Ultrasound Guided Pericapsular Nerve Group Block and Quadratus Lumborum Block for pain relief During patient Positioning for Spinal Anesthesia in proximal femur fracture surgeries. A total of 42 patients enrolled and randomly assigned to either the PENG or QLB group (n=21 each). pain relief will be assessed using the visual analog scale (VAS) at rest and during movement before and after the block, as well as the time of first rescue analgesia and total analgesic consumption. the study will also evaluate the ease of spinal positioning and anesthesiologist satisfaction. patient will be monitored intraoperatively and postoperatively for pain scores. adverse events, and analgesic requirement.

DETAILED DESCRIPTION:
The study aim to compare between ultrasound guided pericapsular nerve group block ( PENG) and quadratus lumborum (QLB) block using VAS score to assess the overall efficacy for pain relief during patient positioning for spinal anesthesia.

After approval of anesthesiology department scientific and ethical committees in Ain Shams University Hospitals, 42 patients will be included in the study, and will be divided into two groups (n=21; each); group PENG and QLB group.

The two groups will be adequately monitored and assessed before spinal anesthesia and post-operatively and they will be compared regarding analgesic outcome by using the visual analogue scaling system, besides, recording time for first call for rescue analgesia and total amount of analgesia require.

Preoperative setting:

Complete history taking and full physical examination. Routine preoperative investigations will be done to all patients including laboratory investigations (complete blood picture, liver function tests, prothrombin time and partial thromboplastin time) and other as needed by the patient condition ( e.g. kidney function, ECHO, ECG, chest X-ray Written informed consent will be obtained from all participants prior to the study.

In the preoperative room: pain score at rest (VAS-R) and at 15-degree passive limb elevation in the supine position to assess pain during movement (dynamic VAS (VAS-D)) will be recorded before giving block.

The two blocks will be performed by the most experienced anesthesiologist in the group.

In group A (PENG): the regional block will be performed with the patient in the supine position. Ultrasound machine with low frequency curvilinear probe (2-5MHz) covered with sterile sheath (Sonoscape® SSI 6000, China) will be initially placed in a transverse plane over the Anterior Inferior Iliac Spine (AIIS) and then aligned with the pubic ramus by rotating the probe counter-clockwise approximately 45 degrees. In this view, the Iliopectineal Eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A 22-gauge, 80-mm needle (B- Braun Medical Inc., Bethlehem, PA, USA) will be inserted from lateral to medial to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution (30ml of bupivacaine 0.25%) will be injected in 5-mL increments while observing for adequate fluid spread in this plane, without exceeding the toxic dose (3 mg/kg).

In group B (QLB): the block will be performed with the patient in the supine position. Under ultrasound guidance with a low frequency curvilinear probe (2-5MHz) covered with sterile sheath (Sonoscape® SSI 6000, China), the probe will be placed in coronal plane at midaxillary line between subcostal margin and iliac crest. A 22-gauge, 80-mm needle (B- Braun Medical Inc., Bethlehem, PA, USA) will be inserted distal to subcostal margin and advanced under curvilinear probe. The needle will be advanced through external oblique aponeurosis, internal oblique, and transversus abdominis muscles. Visualizing the tip penetrating the posterior epimysium of QLM and entering anterior thoracolumbar fascia (ATLF). A small volume of local anesthetic will be injected after locating the needle tip and a negative aspiration for blood. After the distribution of the local anesthetic will be seen, the rest of the 30 mL of 0.25 % of bupivacaine will be injected.

Following the block, heart rate and mean blood pressure will be recorded every 5 min to ensure the blockade is adequate and to monitor the sign of local anesthetic toxicity for 15 min.

If local anesthetic toxicity occurred, cardiovascular and respiratory support and 20% intralipid bolus of 1.5 ml/kg over 2-3 min will be given.

VAS will be assessed at rest (VAS-R) and 15-degree limb elevation (VAS-D) every 10 min for 30 min. After 30 min, patients will be shifted to the operative room.

The median reduction in the VAS score from baseline to 30 minutes will be recorded.

Intraoperative setting:

An intravenous ringer lactate infusion (10-20 ml/kg for 15-20 minutes ) prior to the administration of spinal anesthesia. The patient will be monitored during the procedure using pulse oximetry, non-invasive blood pressure and electrocardiogram.

Patients will be asked to sit for spinal anesthesia. At that time, comfort during sitting for spinal anesthesia will be assessed by the ease of spinal position score (EOSP) (1-sitting without pain and minimal help, 2-mild pain detected by grimacing or verbal expression, 3-severe pain but tolerates positioning with help, 4-unable to sit, requires additional analgesia) . The anesthesiologist who perform spinal anesthesia will be surveyed by team members for operator satisfaction (excellent, good, average, poor) regarding the patient's position. If the patient cannot sit due to pain and VAS was ≥ 4, it will be considered block failure. The patient will be excluded from the study, then patient will receive general anesthesia.

All patients will receive the standard technique of spinal anesthesia in the sitting position after 30 min from the performance of the block by an expert anesthesiologist who is blind and different from the anesthesiologist who perform the two blocks.

For the two groups, spinal anesthesia will be performed under complete aseptic conditions using spinal needle of 25-G, 3 ml bupivacaine 0.5% (heavy Marcaine). Intraoperative antiemetic will be routinely administered, in form of dexamethasone 8 mg IV and ondansetron 4 mg I.V unless contraindicated.

The VAS score will be measured immediately postoperatively and every 2 hours during the first 6 hours and then every 6 hours for only first 24 hours postoperative while patients still at hospital.

If the VAS score is > 4, rescue analgesia will be given; a nalbuphine 0.2 mg/kg IV ; first analgesic request time and the total dose of nalbuphine will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging > 21 years of both sexes.
* Patients scheduled for fixation of proximal femur fracture under spinal anesthesia.
* ASA Physical Status Class I, II or ш.

Exclusion Criteria:

* Patient refusal to participate.
* Patients receiving opioids for chronic analgesic therapy.
* in ability to comprehend the visual analog scale.
* Coagulopathy ( INR > 1.4, platelets < 80000/mm3, or bleeding disorder).
* Infection at the injection site.
* Allergy to local anesthetics.
* Polytroma patients ( e.g., concurrent major thoracic/ abdominal injuries)
* Severe cardiopulmonary disease (e.g., low fixed cardiac output, NYHA class 3/4).
* Neurological disease (e.g., peripheral neuropathy, multiple sclerosis).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
difference in dynamic visual analog scale (VAS - D) scores at 30 minutes post. - block | baseline ( pre - block ) to 30 minutes post block.
  comparison of median reduction in VAS - D scores ( during 15 - degree limb elevation ) between ultrasound - guided pericapsular nerve group block and quadratus lumborum block at 30 minutes after block administration.
  scale: VAS ( 0 - 10 cm; 0 = no pain, 10 = worst pain )

SECONDARY OUTCOMES:
ease of spinal positioning score (EOSP) | immediately before spinal anesthesia ( 30 minutes post - block )
  assessed during sitting for spinal anesthesia using a 4 - point ordinal scale
  1. sitting without pain and minimal help.
  2. mild pain detected by grimacing or verbal expression.
  3. severe pain but tolerates positioning with help.
  4. unable to sit, requires additional analgesia)
operator satisfaction score | immediately after spinal anesthesia placement.
  rated by the anesthesiologist preforming spinal anesthesia on a 4 - point scale: excellent, good, average, poor
postoperative pain score | first 24 hours post - surgery
  visual analog scale score recorded at: 0 hour postoperative, 2 hour, 4 hour, 6 hour, 12 hour and 24 hour postoperatively.
time of first rescue analgesia | up to 24 hours post - block
  time ( minutes ) from block administration to first request for rescue analgesia ( nalbuphine )
total rescue analgesia consumption | first 24 hours post - surgery
  cumulative dose of nalbuphine ( mg ) administered in the first 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Abassya, Egypt